CLINICAL TRIAL: NCT00592982
Title: Bisphosphonate-Associated Jaw Osteonecrosis and PET Imaging
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 73319
Record Dates: First submitted 2007-12-27; First posted 2008-01-14 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Bisphosphonate-associated ONJ; Osteomyelitis of the Jaw; Osteolytic Lesions of the Jaw; Osteoradionecrosis of the Jaw

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. Bisphosphonate-associated osteonecrosis of the jaw(ONJ)is detectable by positron emission tomography(PET).
2. Bisphosphonate-associated ONJ can be diagnosed and characteristically differentiated from other bony pathologies of the jaw(osteomyelitis, osteolytic lesions, and osteoradionecrosis)by PET imaging.

DETAILED DESCRIPTION:
Is to review medical records of approximately 1000 patients with bisphosphonate-associated ONJ who have had PET imaging at the time of diagnosis. Also to review medical records of patients who have been diagnosed with jaw osteomyelitis, osteoradionecrosis, and cancerous lytic lesions who received PET imaging at the time of diagnosis.

If sufficient information regarding presentation and treatment cannot be obtained form the medical record, approximately 300 patients will contacted by mail (and phone if necessary) by the PI or sub-investigators to question them regarding the onset of symptoms, treatment interventions, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bisphosphonate-associated ONJ, osteomyelitis, osteoradionecrosis,and osteolytic lesions who received PET imaging at presentation

Exclusion Criteria:

* Anyone who has not been diagnosed with bisphosphonate-associated ONJ, osteomyelitis, osteoradionecrosis,or osteolytic lesions who received PET imaging at presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Stack, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] 1. Osteonecrosis of the Jaw and Bisphosphonates 2005. NEJM 353: 99-102. 2. Marx RE. 2003 Pamidronate (AREDIA) and Zoledronate (ZOMETA) induced avascular necrosis of the jaws: a growing epidemic J Oral Maxillofac Surg 61:1115-1118 3. Hellstein JW, Marek CL. 2005. Bisphosphonate Osteochemonecrosis (Bis-Phossy Jaw): Is This Phossy Jaw of the 21st Century? J Oral Maxillofac Surg 63: 682-689. 4. Ruggiero SL, Mehrotra B, Rosenberg TJ, Engroff SL. 2004. Osteonecrosis of the Jaws Associated With the Use of Bisphosphonates: A Review of 63 Cases. J Oral Maxillofac Surg 62:527-534. 5. Clarke BM, Boyette JR, Vural EA, Suen JY, Anaisse EJ, Stack BC. Bisphosphonates and Jaw Osteonecrosis: Our Experience. Otolaryngol Head Neck Surg. 2007 Mar;136(3):396-400.